CLINICAL TRIAL: NCT03270254
Title: A Split-mouth Randomised Controlled Clinical Trial of Photodynamic Therapy (PDT) as Adjunctive Therapy to Root Surface Debridement (RSD), Compared to RSD Alone in the Treatment of Residual Periodontal Pockets in Patients With Chronic Periodontitis
Brief Title: Photodynamic Therapy Plus Root Debridement in Gum Disease Treatment V2
Acronym: PDTV2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Ondine Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STH19404
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomised Split mouth
Who Masked: Outcomes Assessor
Masking Description: The patient and Dentist will both be aware of the type of treatment, The researcher analysing the collected samples will be blind to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- root surface debridement (RSD) (No Intervention): Standard care - root surface debridement (RSD)
- light activated dye (PDT) (Active Comparator): light activated dye photodynamic therapy (PDT)
  Interventions: Device: light activated dye photodynamic therapy (PDT)

INTERVENTIONS:
Device: light activated dye photodynamic therapy (PDT) — light activated dye photodynamic therapy-PDT to periodontal pockets
  Arms: light activated dye (PDT)

SUMMARY:
Gum disease is a common disease, which affects 45% of the UK adult dentate population. It is caused by bacteria in dental plaque, which produces inflammation and a deepening of the natural crevice between the gum and the tooth surface. A crevice of 3mm is considered to be within the normal range, but anything ≥4mm is considered to be abnormal and is called a "pocket". Standard treatment of gum disease is mechanical cleaning aimed at removing bacteria off the root surfaces of the teeth. For most teeth, in the majority of patients, this can be achieved by root surface debridement (RSD), which involves passing instruments into the gum pockets to clean the roots. Previous studies have shown that the outcome of treatment is less effective when the pockets are deeper, or where there is bone or root anatomy which makes access for RSD difficult. In such instances additional approaches, such as repeating RSD, surgical access, or the additional use of antibiotics are considered. This clinical study will investigate the benefits and drawbacks of using a light source and dye (photodynamic therapy - PDT) as an additional treatment compared to the standard treatment of RSD alone. Patients with chronic gum problems who have undergone 1 cycle of RSD, but have residual pockets will be invited to join the study. All residual pockets will be treated with the conventional treatment of RSD. Following a random allocation process the residual pockets in half the mouth will receive additional treatment with PDT at the same appointment. Patients will be followed up for 3 months to evaluate the clinical benefits and any side effects. The aim of the study is therefore to evaluate if this localised, simple treatment can add benefit to RSD alone, thus reducing the need for antibiotics or surgery to treat residual pockets.

DETAILED DESCRIPTION:
The study will be a single centre, examiner masked, two arm, split mouth, randomized controlled clinical trial, to evaluate the clinical effectiveness of mechanical cleaning (RSD) plus additional use of a light activated dye (photodynamic therapy-PDT) compared to mechanical cleaning alone, in the treatment of residual pockets, in patients with chronic gum disease. The null hypothesis is that there is no difference between RSD and the additional use of PDT compared to RSD alone, when treating patients with chronic gum disease. The local delivery treatment of PDT requires the low power light to be shone into the pocket for 1 minute in order to activate the dye which kills the bacteria. For this reason it is a treatment which is more suited to treating localised rather than widespread disease. Thus, patients with chronic gum problems who have had a cycle of treatment with the hygienist, but have a few residual pockets will be selected for this study. Subjects will be recruited from patients attending the hygienist following a first cycle of RSD, who have sufficient remaining disease to represent a meaningful challenge. This reflects the normal care pathway for patients, where simple approaches to treatment are followed up with more complicated therapy for any areas which fail to respond. A power calculation has shown that 29 patients are expected to be enough to see if PDT & RSD can produce better gum health than RSD alone. However, to account for unexpected patient withdrawals, 35 patients will be recruited to this study. The staff hygienists in the department are capable of providing treatment for 60-90 patients over a 3-month period. Out of these patients those with more severe disease are likely to have residual pockets that require further cycles of RSD. Thus there is potentially a good population of patients attending Charles Clifford Dental Hospital to recruit from. All residual sites within a subject who participates in the study will be treated by mechanical cleaning. This is the standard treatment which would apply for most patients in this situation. A random allocation procedure will be used to designate sections of the mouth to receive additional treatment with the PDT. This will not be made known to the operator performing the RSD until after they have completed that aspect of treatment. This helps reduce bias as the operator will clean all sites to an equivalent standard. The split mouth approach means that the patient will act as their own control. This helps reduce the numbers of patients which need to be recruited as compared to a study with 2 parallel groups, where each group receives a different treatment. The suggested disadvantage of a split mouth design, is the fact that there may be some contamination of RSD sites only with the action of a chemical remote from the site it was originally placed in. However, in this study the chemical needs to be activated by the light, and therefore it is easier to control the activity of PDT therapy to the sites it was designated to be used in. For this reason there needs to be a gap between the section of the mouth treated by adjunctive PDT & RSD, compared to the section of the mouth where RSD alone is the treatment. No additional appointments will be required of the patients compared to the normal protocol as they will receive the "gold standard" treatment of mechanical cleaning (RSD) in all sites. The additional requirements of the study will be the time it takes to provide treatment using PDT. This is anticipated to be between 5-15 minutes depending upon the number and distribution of sites throughout the mouth. Sample collection of bacterial plaque and gum fluid from 2 sites per patient will take an additional 5-10 minutes. The normal treatment time at this stage of treatment would be 60 minutes and this will be extended to 70-85 minutes for the study purposes. None of the additional procedures are likely to cause discomfort. The 3 month re-assessment examination will require repeat sample collection of bacterial plaque and gum fluid from 2 sites which will take an additional 5-10 minutes. Thus the standard patient reassessment appointment of 60 minutes will be extended to 65-70 minutes. The full process from recruitment of patients to writing up this student project is expected to be finished within seven to nine months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 30 years old
* Presence of at least 20 remaining teeth
* Patients diagnosed with moderate to severe chronic periodontitis, according to Armitage 1999 classification
* Have undergone a minimum of one cycle of full mouth nonsurgical root surface debridement.
* A minimum of 8 residual periodontal pockets (≥4mm) per patient and a maximum of 24. Amongst these, at least one site per half mouth must exhibit pocket depths of ≥ 6 mm.
* Pockets distribution should allow for split mouth design using sextants in a diagonal orientation.
* Received no active periodontal treatment for the last three months.
* Full mouth plaque score and full mouth bleeding score ≤ 30%.
* Sites in the other half of the mouth to be separated by one or more teeth (avoids photosensitising agent affecting the other half).

Exclusion Criteria:

* Patients with systemic diseases that may alter the response to treatment and healing in periodontal diseases.
* Pregnancy and lactation.
* The use of systemic or local antibiotic in the past three months.
* The need for antibiotic prophylaxis before periodontal treatment.
* Use of antimicrobial mouth rinses in the preceding two months.
* The use of any pharmacological agents that could influence the study outcome or inflammatory indicators (e.g. patients currently on photosensitizing medications).
* Confirmed or suspected allergy or hypersensitivity to methylene blue.
* Confirmed or suspected allergy or hypersensitivity to chlorhexidine.
* Confirmed or suspected allergy or hypersensitivity to polymethyl methacrylate (PMMA).
* Patients with severe glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Inability to perform proper oral hygiene due to physical impairment.
* Patients unable to consent for themselves.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Pocket depth change | 3 months
  The difference in mean change of probing pocket depth in millimetres between the test and control sites

SECONDARY OUTCOMES:
Change in clinical attachment | 3 months
  The difference in mean change of clinical attachment loss in millimetres between the test and control sites.
Bleeding on probing | 3 months
  The percentage difference of bleeding on probing between tests and controls.
Probing depths originally ≥ 6mm. | 3 months
  The percentage difference of sites with probing depths originally ≥ 6mm.
Probing depths originally ≤3mm | 3 months
  The percentage increase of sites with probing depths originally ≤3mm
Number of sites improving by ≥2mm | 3 months
  The total number of sites improving by ≥2mm
Percentage of sites improving by ≥2mm | 3 months
  The percentage of sites improving by ≥2mm

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Griffiths, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The research findings will probably be published in a scientific journal